CLINICAL TRIAL: NCT02560324
Title: Repurposing Melatonin Receptor Agonists as Adjunct Treatments for Smoking Cessation
Brief Title: Effect of Ramelteon on Smoking Abstinence
Acronym: RAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 823286; R21DA040902 (NIH)
Record Dates: First submitted 2015-09-23; First posted 2015-09-25 (Estimated); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-11

CONDITIONS: Tobacco Use Disorder
Keywords: Ramelteon; Nicotine; Nicotine dependence; Insomnia; Tobacco Dependence
MeSH Terms: conditions — Tobacco Use Disorder; Sleep Initiation and Maintenance Disorders | interventions — ramelteon; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ramelteon (Experimental): The study will be performed using 8mg of ramelteon, which is currently marketed for the treatment of sleep problems. The proposed study follows the typical dosing regimen for ramelteon (8mg once a day) for 5 days during each quit assessment period.
  Ramelteon will be purchased and packaged into blister packs by the Investigational Drug Service (IDS) at the University of Pennsylvania. In accordance with FDA recommendations, subjects will be instructed to take study medication within 30 min prior to going to bed and avoid taking study medication with or immediately after a high fat meal.
  Interventions: Drug: Ramelteon
- Placebo (Placebo Comparator): 5-day placebo-controlled medication period.
  Placebo ingredients will be purchased, encapsulated, and packaged into blister packs by the IDS at UPenn. Both active medication and placebo will look identical.
  The study medication assignments for each participant in this project is randomized and counterbalanced. This means that approximately 50% of participants will take ramelteon during the first medication period, followed by the placebo in the second medication period. Alternatively, approximately 50% of participants will take the placebo during the first medication period, followed by ramelteon during the second medication period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon
  Arms: Ramelteon
Drug: Placebo
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled crossover study to test whether a medication called ramelteon (Brand Name: Remeron) will help smokers quit and whether it reduces sleep problems that smokers experience during a quit attempt.

DETAILED DESCRIPTION:
Ramelteon, an FDA-approved treatment for insomnia, is used to treat sleep problems (e.g., specifically sleep onset latency) by enhancing melatonin receptor function. The investigators propose a randomized double-blind placebo-controlled crossover study.

Fifty chronic smokers will complete a validated procedure for screening new medications. All subjects will receive 8mg ramelteon and placebo. The order in which ramelteon and placebo is received will be randomized across participants. This is a 6-week study consisting of two 2-week medication phases separated by a 2-week washout. Each phase includes 1 week of ad libitum smoking (baseline) and 1 week of medication (ramelteon vs. placebo) plus transdermal nicotine patches while trying to abstain from smoking (quit assessment). Subjects will complete the same procedures during each study phase. Following completion of the study, participants will be offered standard smoking cessation treatment.

For the duration of the study, subjects will be asked to keep sleep diaries and to wear an armband while sleeping, which provides objective indices of sleep duration and quality (SensewearPro® armband).

The primary outcome will be the total number of days abstinent (out of 5) during each quit assessment period. Intermediate outcomes include sleep onset latency (self-report) and sleep efficiency (SensewearPro®).

This study will provide information about the role of the melatonin system during brief abstinence and whether enhancing melatonin reduces abstinence-induced sleep problems that promote smoking relapse. Information obtained in this study may further establish the role of sleep disturbance in promoting smoking relapse.

ELIGIBILITY:
Inclusion Criteria:

1. Smokers who are between 18 and 65 years of age who self-report smoking at least 10 cigarettes per day for at least the last 6 months.
2. Interest in quitting smoking in the next 2 to 4 months.
3. Healthy as determined by the Study Physician, based on a medical evaluation including medical history and physical examination, and psychiatric evaluation.
4. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent and HIPAA form.
5. Women of childbearing potential must consent to use a medically accepted method of birth control while participating in the study (e.g., condoms and spermicide, oral contraceptive, Depo-provera injection, contraceptive patch, tubal ligation).

Exclusion Criteria:

Smoking Behavior:

1. Current enrollment in a smoking cessation program, or use of other smoking cessation medications in the last month or plans to do either in the next 2 months.
2. Daily use of chewing tobacco, snuff and/or snus, or electronic cigarettes.
3. Provide a carbon monoxide (CO) breath sample reading less than 10 parts per million (ppm) at Intake.

Alcohol/Drugs:

1. Self-report current alcohol consumption that exceeds 25 standard drinks/week over the past 6 months. Subjects will be told to limit or avoid the use of alcohol while in the study to avoid any adverse reactions to the study medication.
2. Self-reports substance use disorders (abuse or dependence involving alcohol, opiates, cocaine or other stimulants, or benzodiazepines; not nicotine) in the last 6 months.
3. Providing a breath alcohol concentration (BrAC) reading of greater than or equal to 0.01 during any session.
4. A positive urine drug screen for cocaine, amphetamines, methamphetamines, benzodiazepines, PCP, methadone, barbiturates, marijuana, ecstasy (MDMA), oxycodone, tricyclic antidepressants, and opiates (low level cut-off 300 ng/mL) during any session.

Psychiatric Exclusion (as determined by self-report on phone screen and/or through MINI during Intake):

1. Current psychiatric disorders (depression, bipolar, schizophrenia, hypomanic/manic episode) as determined by self-report and/or MINI psychological interview.
2. Past history of psychiatric disorders (including suicide attempt) other than depression as determined by self-report and/or MINI psychological interview.
3. Suicide risk score on MINI greater than 1.

Medical:

1. Females who are currently pregnant, planning a pregnancy during the study, or currently breastfeeding/lactating. All female subjects shall undergo a urine pregnancy test at the Intake and must agree in writing to use an approved method of contraception. Following enrollment, pregnancy tests will be conducted at the beginning of each baseline week.
2. For those with a history of jaundice/liver disease: liver function tests more than 20% outside of the normal range; Gamma-glutamyl Transpepsidase (GGT) values more than 20% outside of the normal range. If Albumin/Globulin ratios are 20% outside of normal range the abnormal value will be evaluated for clinical significance by the Study Physician and eligibility will determined on a case-by-case basis.
3. Heart/Cardiovascular disease (e.g., angina, coronary heart disease, stroke, etc.) in the past 6 months.
4. Endocrine or metabolic disorders (e.g., Type-I diabetes).
5. Blood disorders (e.g., anemia or hemophilia).
6. Uncontrolled hypertension (BP systolic greater than 159 and/or diastolic greater than 99)*.
7. Clinically significant dyssomnia (except insomnia; e.g. sleep apnea syndrome, narcolepsy).

   * Participants presenting with SBP greater than 159 mmHg and/or DBP greater than 99 mmHg at the Intake visit will be instructed to sit quietly for 10 minutes. Then the participant will have a second blood pressure reading taken after a 10 minute period. If, after the second reading the SBP greater than 159 mmHg and the DBP greater than 99 mmHg, the individual will be instructed to sit comfortably for 10 minutes and then have a third blood pressure reading. If, after the third reading the SBP greater than 159 mmHg and the DBP greater than 99 mmHg, the individual will be ineligible to participate.

Medication:

1. Current use or recent discontinuation (within the past month) of any of the following medications:

   1. Anti-anxiety or panic disorder medications (e.g., clonazepam, alprazolam).
   2. Anti-psychotic medications (e.g., thorazine, Seroquel).
   3. Mood-stabilizers (e.g., Lithium, Lamictal/lamotrigine, valproic acid, Neurontin/gabapentin, Topamax/topiramate, Tegretol/carbamazepine).
   4. Prescription stimulants (e.g., Provigil, Ritalin, Adderall).
   5. Medications contraindicated with ramelteon (e.g., fluvoxamine, buprenorphine or other medications metabolized by certain cytochrome P450 enzymes)
2. Current use or recent discontinuation (within the past 2 weeks) of any of the following medications (subjects must agree to refrain from using any other sleep aids while enrolled in the study):

   1. Sleep medications (e.g., zolpidem/Ambien, eszopiclone/Lunesta)
   2. Over-the-counter sleep aids (e.g., melatonin, diphenhydramine/Benadryl)
3. Daily use of opiate-containing medications for chronic pain (Duragesic/fentanyl patches, Percocet, Oxycontin). Smokers who report taking opiate-containing medications on an "as-needed" basis will be instructed to refrain from use until their study participation is over and that they will be tested to ensure they have complied with this requirement.
4. Known allergy to study medication (e.g., angioedema).

Subjects will be instructed to refrain from using any study prohibited drugs/medications (both recreational and prescription) throughout their participation in the study. After final eligibility is confirmed, subjects who report taking contraindicated medication(s) over the course of the study period may only remain eligible if the Study Physician and/or Principal Investigator determines that the contraindicated medication(s) do/did not impact the study design, data quality, and/or subject safety/welfare. Subjects are permitted to take necessary prescription medications not included within the exclusion list during the study.

General Exclusion:

1. Current, anticipated, or pending enrollment in another research program over the next 2-3 months that could potentially affect subject safety and/or the study data/design as determined by the Principal Investigator and/or Study Physician.
2. Not planning to live in the area for the next two months.
3. Currently working night shift or rotating shift or other habitual alteration of the sleep/wake cycle.
4. Allergy to latex or adhesive tape.
5. Inability to provide informed consent or complete any of the study tasks as determined by the Principal Investigator.
6. Not able to effectively communicate in English (reading, writing, speaking).
7. Missing 2 or more doses during the medication period determined by self-report.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Ashare, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Interdisciplinary Research on Nicotine Addiction, School of Medicine, University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 697 potential participants were pre-screened over the phone for eligibility between September 2015 and August 2018. 140 potential participants attended an in-person eligibility screen at the research clinic.
Pre-assignment Details: 69 of 140 participants met eligibility criteria and were randomized. For participants who were not randomized: 61 did not meet inclusion criteria, 5 declined to participate, 4 missed the baseline visit, and 1 is unknown.
Groups:
- Ramelteon Then Placebo: Participants smoked ad libitum for 1 week and then received 8mg of Ramelteon once per day + transdermal nicotine for 1 week. After a washout period of 2 weeks, participants again smoked ad libitum for 1 week, then received Placebo pills (matching Ramelteon 8mg pills) once per day + transdermal nicotine for 1 week.
- Placebo Then Ramelteon: Participants smoked ad libitum for 1 week and then received Placebo pills (matching Ramelteon 8mg pills) once per day + transdermal nicotine for 1 week. After a washout period of 2 weeks, participants again smoked ad libitum for 1 week, then received 8mg of Ramelteon once per day + transdermal nicotine for 1 week.
Period: Period 1 (2 Weeks)
Arm/Group | Ramelteon Then Placebo | Placebo Then Ramelteon
Started | 35 | 34
Completed | 23 | 25
Not Completed | 12 | 9
Period: Washout (2 Weeks)
Arm/Group | Ramelteon Then Placebo | Placebo Then Ramelteon
Started | 23 | 25
Completed | 23 | 23
Not Completed | 0 | 2
Period: Period 2 (2 Weeks)
Arm/Group | Ramelteon Then Placebo | Placebo Then Ramelteon
Started | 23 | 23
Completed | 22 | 21
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ramelteon Then Placebo | Placebo Then Ramelteon | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (8.9) | 52.1 (7.4) | 50 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 16 | 11 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 15 | 16 | 31
  White | 6 | 5 | 11
  More than one race | 1 | 0 | 1
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes smoked per day] | 12.1 (3.3) | 16.6 (8.4) | 14.3 (6.7)
Education [Count of Participants; unit: Participants]
  HS/GED or less | 9 | 13 | 22
  Some college or more | 13 | 8 | 21
Income [Count of Participants; unit: Participants]
  < $20,000 | 16 | 13 | 29
  > $20,000 | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Smoke-free Days (Biochemically Verified) During Each 5-day Quit Assessment.
Description: The quit assessment will begin the Monday morning of each quit week and will end that Friday. The total number of days of abstinence will be assessed.
Time Frame: Week 2 and Week 6
Measure: Mean (Standard Deviation); unit: days of smoking abstinence
Groups:
- Ramelteon: Participants received 8mg of Ramelteon once per day + transdermal nicotine for 1 week.
- Placebo: Participants received Placebo pills (matching Ramelteon 8mg pills) once per day + transdermal nicotine for 1 week.
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 43 | 43
days of smoking abstinence | 2.7 (1.6) | 2.6 (1.6)

2. Secondary Outcome: Subjective Sleep Disturbance
Description: Sleep onset latency will be assessed via daily sleep diaries during each quit assessment.
Time Frame: Week 2 and Week 6
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 43 | 43
minutes | 20.8 (12.7) | 23.7 (23.9)

3. Secondary Outcome: Objective Sleep Disturbance
Description: Sleep efficiency (% of time in bed spent sleeping) will be assessed via the SensewearPro armbands during each quit assessment.
Time Frame: Week 2 and Week 6
Measure: Mean (Standard Deviation); unit: % of time in bed spent sleeping
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 43 | 43
% of time in bed spent sleeping | 86.7 (12.5) | 86.6 (12.5)

4. Secondary Outcome: Side Effects of Ramelteon
Description: Side effects will be assessed at each in-person visit using a Side Effects Checklist (SEC) that lists 21 possible side effects of ramelteon. The scale for rating each side effect is None=0, Mild=1, Moderate=2, and Severe=3. The higher the score, the more side effects reported by the participant. The minimum score is 0 and the maximum score is 3 for each possible item on the scale. The Outcome Measure is an average of the 21 listed side effects.
Time Frame: Baseline (weeks 1 and 5); Quit assessments (weeks 2 and 6)
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Ramelteon (Baseline): Before participants received 8mg of Ramelteon once per day + transdermal nicotine for 1 week.
- Placebo (Baseline): Before participants received Placebo pills (matching Ramelteon 8mg pills) once per day + transdermal nicotine for 1 week.
- Ramelteon (Quit Week): Participants received 8mg of Ramelteon once per day + transdermal nicotine for 1 week.
- Placebo (Quit Week): Participants received Placebo pills (matching Ramelteon 8mg pills) once per day + transdermal nicotine for 1 week.
Arm/Group | Ramelteon (Baseline) | Placebo (Baseline) | Ramelteon (Quit Week) | Placebo (Quit Week)
Number analyzed (Participants) | 43 | 43 | 43 | 43
scores on a scale | 0.028 (0.057) | 0.034 (0.047) | 0.05 (0.078) | 0.027 (0.041)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 7 weeks
Groups:
- Ramelteon: Participants received medication (8mg of Ramelteon) once per day + transdermal nicotine for 1 week.
- Placebo: Participants received Placebo once per day + transdermal nicotine for 1 week.
Arm/Group | Ramelteon | Placebo
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/57
Other Adverse Events (participants affected / at risk) | 22/58 | 21/57
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramelteon (N=58) | Placebo (N=57)
Headache (Nervous system disorders) | 11 (21) | 12 (20)
Insomnia/Trouble Sleeping (General disorders) | 12 (34) | 9 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/24/NCT02560324/Prot_SAP_000.pdf